CLINICAL TRIAL: NCT00814697
Title: Open-label, Exploratory Study of the Efficacy of Repetitive Transcranial Magnetic Stimulation on Naming and Verbal Fluency in Patients With Alzheimer's Disease With Functional Imaging Correlates
Brief Title: Effect of Repetitive Transcranial Magnetic Stimulation on Language in Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The New York Memory Services (Other)
Responsible Party: Principal Investigator, Gayatri Devi, MD, Clinical Associate Professor of Neurology & Psychiatry, The New York Memory Services
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 91913-5
Record Dates: First submitted 2008-12-24; First posted 2008-12-25 (Estimated); Results first posted 2014-01-28 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Alzheimer's Disease; Aphasia; Dementia
Keywords: Alzheimer; Language; Treatment; TMS; rTMS
MeSH Terms: conditions — Alzheimer Disease; Aphasia; Dementia; Language

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transcranial Magnetic Stimulation (Experimental): Repetitive Transcranial Magnetic Coil Stimulation (rTMS) treatment in Alzheimer's disease. The Magstim Rapid2 stimulator with a peak magnetic field of 0.5-3.5 Tesla at 100% output was used over the right and left dorsolateral prefrontal cortex. Patients received 4 sessions of rTMS over 2 weeks, lasting approximately 30 minutes, 2 consecutive days a week for 2 weeks.
  Interventions: Device: Repetitive Transcranial Magnetic Coil Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Coil Stimulation (rTMS) — The first six patients were administered rTMS at 10Hz in 20 trains of 5 seconds with 20 second intervals between trains in each hemisphere. The total number of pulses for each session was set at 1000 pulses. The second six enrolled patients were administered rTMS at 15 Hz in 20 trains of 5 seconds with 25 second intervals between trains in each hemisphere.

SUMMARY:
The investigators wish to investigate the efficacy of targeted repetitive transcranial magnetic stimulation (rTMS) on expressive language in patients with Alzheimer's disease (AD). In rTMS, magnetic pulses are used to noninvasively stimulate focal areas of cortex of about a square centimeter in area. rTMS has been approved in the United States for the diagnosis of peripheral nerve conditions.

Depending on the frequency of stimulation, rTMS can preferentially stimulate or inhibit cortical areas. In stroke rehabilitation, for example, inhibition of the contralateral, uninvolved hemisphere by low frequency rTMS has improved movement of the affected limbs because of less aberrant inhibition of the affected hemisphere by the healthy hemisphere. The effects of rTMS has also been investigated and found to be useful in treating refractory depression and depression in Parkinson's disease. In addition, rTMS has improved naming in patients with Alzheimer's disease and has improved cognitive abilities and memory in non-demented older adults. Two studies found that rTMS improved aphasia in patients with stroke. While these studies are small, a review of the literature suggests that there may be a beneficial role for rTMS in patients with chronic neurological conditions. In addition, rTMS appears to be well tolerated, with transient headaches being the most common side effect.

In this small open label study, the investigators wish to investigate the usefulness of bilateral stimulation of the brain region termed the dorsolateral prefrontal cortex (DLPFC) in patients with AD who have naming and language deficits.

DETAILED DESCRIPTION:
Subjects for this study will be recruited from Dr. Devi's clinical practice. Eligible subjects must have a diagnosis of possible or probable Alzheimer's disease using NINCDS-ADRDA criteria. The patient and his or her legally authorized representative need to be available to sign the informed consent. The assent of the incapable subject will be obtained prior to enrolling the subject in the study.

Once informed consent and assent are obtained, the subject will have a functional magnetic resonance imaging (fMRI) scan of their brain anytime during the 2 weeks prior to the first study visit. At Visit 1, subjects will undergo a baseline battery of cognitive tests lasting approximately 30 minutes. Subsequently, the subject will undergo rTMS.

During the visit, Dr. Devi will locate the area of the brain to be stimulated and mark that area of the scalp with an indelible skin marker that will wash out over time. In addition, the subjects will be provided with ear plugs to use during stimulation. This process of locating the area to be stimulated will take about an hour and will occur once. Then rTMS will be started and this procedure will take approximately 20-30 minutes (please see the full protocol for a complete description of this process).

Each rTMS stimulation session will last for about 30 minutes, 2 consecutive days a week for 2 weeks. Both immediately prior to the onset of the first rTMS session, and just after the end of the fourth and final rTMS session, subjects will be tested on their cognitive and language skills. These two testing sessions will last 30 minutes each. Subjects will have another fMRI scan anytime during the 2 days after the fourth and final rTMS stimulation session.

Subjects will continue to receive usual care throughout the study period. Any changes to usual treatment will be noted in the study file.

All subjects will be seen again 4 weeks after the final study treatment session and will once again undergo the brief cognitive battery and fMRI scan.

The investigators expect to recruit two subjects at a time for the study and each subject will be enrolled for 5 weeks from the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a diagnosis of probable or possible Alzheimer's disease, diagnosed using standardized criteria.
* If subjects are determined by the PI to lack decisional capacity to consent to the study, a legally authorized representative must be available to sign the informed consent on behalf of the subject. In this case the assent of each subject will be obtained as well. If at any time the subject withdraws his or her assent, the subject will be disenrolled from the study.
* Subjects will score at or below 30 on the 60 item naming section of the Boston Diagnostic Aphasia and/or below 50% on the Controlled Word Association (CFL) Category Naming.

Exclusion Criteria:

* Subjects newly diagnosed with AD and not yet receiving usual care are not eligible.
* Subjects must not have pacemakers.
* They must not have a history of implanted metal objects.
* They must not have a history of seizures or epilepsy.
* There must not be any recent history of migraines.
* There must not be any history of uncontrolled depression.
* They must not be on any medications that will significantly lower the seizure threshold.
* Any other medical condition that is judged by the PI to make rTMS unsafe for the subject.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-12; Primary Completion 2011-12 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gayatri Devi, MD, Principal Investigator — The New York Memory Services
Locations (1):
- The NY Memory Services, New York, New York, United States

REFERENCES:
- [Background] Cotelli M, Manenti R, Cappa SF, Geroldi C, Zanetti O, Rossini PM, Miniussi C. Effect of transcranial magnetic stimulation on action naming in patients with Alzheimer disease. Arch Neurol. 2006 Nov;63(11):1602-4. doi: 10.1001/archneur.63.11.1602. PMID 17101829
- [Background] Ahmed MA, Darwish ES, Khedr EM, El Serogy YM, Ali AM. Effects of low versus high frequencies of repetitive transcranial magnetic stimulation on cognitive function and cortical excitability in Alzheimer's dementia. J Neurol. 2012 Jan;259(1):83-92. doi: 10.1007/s00415-011-6128-4. Epub 2011 Jun 14. PMID 21671144
- [Background] Bentwich J, Dobronevsky E, Aichenbaum S, Shorer R, Peretz R, Khaigrekht M, Marton RG, Rabey JM. Beneficial effect of repetitive transcranial magnetic stimulation combined with cognitive training for the treatment of Alzheimer's disease: a proof of concept study. J Neural Transm (Vienna). 2011 Mar;118(3):463-71. doi: 10.1007/s00702-010-0578-1. Epub 2011 Jan 19. PMID 21246222
- [Background] Rabey JM, Dobronevsky E, Aichenbaum S, Gonen O, Marton RG, Khaigrekht M. Repetitive transcranial magnetic stimulation combined with cognitive training is a safe and effective modality for the treatment of Alzheimer's disease: a randomized, double-blind study. J Neural Transm (Vienna). 2013 May;120(5):813-9. doi: 10.1007/s00702-012-0902-z. Epub 2012 Oct 18. PMID 23076723
- [Background] Cotelli M, Manenti R, Cappa SF, Zanetti O, Miniussi C. Transcranial magnetic stimulation improves naming in Alzheimer disease patients at different stages of cognitive decline. Eur J Neurol. 2008 Dec;15(12):1286-92. doi: 10.1111/j.1468-1331.2008.02202.x. PMID 19049544
- [Background] Cotelli M, Calabria M, Manenti R, Rosini S, Zanetti O, Cappa SF, Miniussi C. Improved language performance in Alzheimer disease following brain stimulation. J Neurol Neurosurg Psychiatry. 2011 Jul;82(7):794-7. doi: 10.1136/jnnp.2009.197848. Epub 2010 Jun 23. PMID 20574108

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were recruited from a tertiary memory disorders practice. Patients were diagnosed as having probable or possible Alzheimer's Disease (AD), using the National Institute of Neurological and Communicative Disorders and Stroke and Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria.
Pre-assignment Details: Exclusion criteria included newly diagnosed AD, pacemaker placement, a history of implanted metal object, seizures or epilepsy, a recent history of migraines, uncontrolled depression and those on medications lowering the seizure threshold.
Groups:
- rTMS: rTMS treatment in Alzheimer's disease
  Repetitive Transcranial Magnetic Coil Stimulation (rTMS) : Using rTMS to treat language deficits in Alzheimer's patients
Period: Overall Study
Arm/Group | rTMS
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | rTMS
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.1 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Assessment Task Scores Before, During and After rTMS.
Description: Cognitive assessment tasks - Boston Diagnostic Aphasia Examination (BDAE), CFL Category naming (CFL), Mini-Mental State Examination (MMSE) - were administered and scored according to standard procedures before, during and 4 weeks after rTMS.
  Higher scores are associated with better cognition; No absolute cut-offs were used here as the outcomes were not categorically assessed.
  Total possible score ranges by test, lowest to highest:
  BDAE - 0 to 15 CFL - 0 to 62 MMSE - 0 to 30 Full range data and means presented below represents range of scores at 4-weeks post-rTMS treatments.
Time Frame: 6 weeks
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Cognitive Assessment: rTMS treatment in Alzheimer's disease
  Repetitive Transcranial Magnetic Coil Stimulation (rTMS) : Using rTMS to treat language deficits in Alzheimer's patients
Arm/Group | Cognitive Assessment
Number analyzed (Participants) | 12
units on a scale
  Mini-Mental State Examination (MMSE) | 26.9 (3.80) [19 to 30]
  Boston Diagnostic Aphasia Examination (BDAE) | 13.3 (2.12) [9 to 15]
  CFL Category Fluency | 17.0 (7.03) [8 to 32]

ADVERSE EVENTS:
Arm/Group | rTMS
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No